CLINICAL TRIAL: NCT00486005
Title: Weight Gain Management in Patients With Schizophrenia During Treatment With Olanzapine in Association With Nizatidine
Brief Title: Weight Gain Management in Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7932; F1D-BL-HGLA
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2007-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — olanzapine-fluoxetine combination; Nizatidine

INTERVENTIONS:
Drug: Olanzapine Hydrochloride
Drug: Nizatidine
Drug: Placebo

SUMMARY:
Evaluate the efficacy of nizatidine in reducing/limiting weight gain in patients with schizophrenia who have been under treatment with olanzapine for at least two months and evaluate the treatment effects on the Eating Inventory, BPRS, number of treatment, emergent adverse events, changes in vital signs, laboratory results and extrapyramidal effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients, men or women, with age of 18 to 65 years
* Patients must have schizophrenia that meets disease diagnostic criteria as defined in DSM-IV Sections 295.10, 295.20, 295.30, or 295.90 and not to be in a clinically acute phase, in accordance with the judgment of the investigator
* Patients in use of 5 mg/day and 20 mg/day of olanzapine for a period not less than 2 months and not greater than 6 months and that have increased at least 5% of their corporal weight since the beginning of the treatment with olanzapine.
* The individuals must be trustworthy, and have a level of understanding enough to carry out all the tests and examinations demanded for the protocol, to understand the nature of the study and to have signed the informed consent
* Women with potential to become pregnant must be using a medically acceptable and reliable means of birth control.

Exclusion Criteria:

* Participation in a clinical study of another drug in investigation within a period of 1 month (30 days) before the entrance in the study (Visit 1)
* People who have used clozapine within a period of 12 months before the beginning of the study
* People with diagnosis of diabetes mellitus types I or II without adjusted clinical control or have initiated the medication use for glycemic control in the last 6 months
* DSM-IV substance (except nicotine and caffeine) dependence within the past 30 days
* Current participation in programs of weight loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2003-02; Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of olanzapine associated to nizatidine compared to olanzapine associated to placebo to prevent/control weight gain

SECONDARY OUTCOMES:
Compare the effect of olanzapine with nizatidine or placebo evaluated by the average alteration between the groups in cognitive control of appetite, disinhibition and susceptibility to hunger, variation of weight and total punctuation in BPRS
Compare the security of the association of olanzapine with nizatidine and olanzapine and placebo in relation to laboratory values, vital signs, and incidence of extrapyramidal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rio de Janeiro, Brazil

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com